CLINICAL TRIAL: NCT01976078
Title: Ontogeny of Voriconazole Pharmacokinetics and Metabolism in Children and Adolescents
Brief Title: Development of Voriconazole Pharmacokinetics and Metabolism in Children and Adolescents
Status: Completed | Type: Observational
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Michael Neely, Associate Professor of Pediatrics, Children's Hospital Los Angeles
Other Study IDs: CCI-11-00334; R01HD070996 (NIH)
Record Dates: First submitted 2013-09-18; First posted 2013-11-05 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Pharmacokinetics; Voriconazole
Keywords: Voriconazole; Pharmacokinetics; Ontogeny; Modeling; Bayesian
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Midazolam/Ranitidine/Esomeprazole: All enrolled subjects will have a study pharmacokinetic visit where they will be given the above cocktail of drugs along with their clinically indicated voriconazole dose, followed by blood sampling over the next 12 hours.
  Interventions: Drug: Midazolam/Ranitidine/Esomeprazole

INTERVENTIONS:
Drug: Midazolam/Ranitidine/Esomeprazole — Each of the three drugs will be given at 10% of their usual doses for age/weight.

SUMMARY:
The death rate in children from the invasive fungal infection called aspergillosis is more than 50%. Voriconazole is the first-line therapy for this infection. In a previous publication the investigators have shown a highly significant relationship between voriconazole plasma concentrations and survival. However, voriconazole dosing is currently poorly established, and plasma drug exposure varies between children by 400% or more, even after intravenous dosing. The objective of this study is to investigate the reasons for this variability in voriconazole pharmacokinetics (PK).In two studies, the investigators will enroll 80 children/adolescents receiving oral or intravenous voriconazole, divided by age under 2 years (n=15), and 2-18 years (n=65). From each patient the investigators will collect the following: 1) a blood sample for detection of several genetic changes known to affect drug metabolizing enzyme (DME) activity; 2) up to 9 blood samples after a voriconazole dose for measurement of voriconazole ("PK sampling"); 3) follow-up samples after each PK sampling visit if necessary to adjust the dose so that voriconazole concentrations in the blood are satisfactory (known as therapeutic drug monitoring or TDM). At the time of the voriconazole dose prior to the PK sampling, we will also give single IV or oral (corresponding to the route of voriconazole administration) low doses of esomeprazole (an antacid), midazolam (a sedative), and ranitidine (an antacid) as a cocktail to test or probe DME activity. All of these medications are used commonly in children already. The investigators will estimate DME activity or phenotype using ratios of probe drug metabolite to parent drug concentrations, while simultaneously quantifying the amount of DME genetic material (mRNA) and protein in white blood cells. The investigators will test associations between DME activity, mRNA, protein, voriconazole PK, age, sex, and degree of illness. The investigators will also use a computer program to integrate all these data to develop a comprehensive model that will predict blood concentrations of voriconazole in children of all ages, as well as assist physicians and pharmacists to dose voriconazole more accurately.The total study duration for each subject will be until after the TDM follow up visit, generally about one week.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will be enrolled before their 18th birthday.
2. Participant/parent/legal guardian must be able and willing to provide signed informed consent.
3. Laboratory values obtained within 7 days prior to study entry (obtained for clinical purposes)

   1. Hemoglobin ≥ 7.0 g/dL (transfusion dependence acceptable)
   2. Aspartate aminotransferase (AST) (SGOT), alanine aminotransferase (ALT) (SGPT), and total bilirubin ≤ 5 X upper limit of age-appropriate normal (ULN)
   3. Serum creatinine ≤ 3 X ULN

Exclusion Criteria:

1. Pregnancy
2. Active substance abuse or other psychiatric illness that would prevent adherence to the study protocol. Investigators will not record this information in the screening log, and the information will be obtained from existing documents in the medical record only.
3. Known hypersensitivity or intolerance to study medications
4. Not expected to survive >1 week.
5. Weight < 4.5 kg (blood volume draw limitations)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with an invasive fungal infection
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2015-04-22 (Actual); Study Completion 2015-04-22 (Actual)

PRIMARY OUTCOMES:
Voriconazole steady-state pharmacokinetics | During the 12 hours after a dose
  8 (after intravenous dosing) or 9 (after oral dosing) samples are taken after a voriconazole dose over a 12 hour timeframe.

SECONDARY OUTCOMES:
Voriconazole drug metabolizing enzyme activity | Within 12 hours after a study medication dosing
  At the time of the voriconazole dose used for the primary outcome, an intravenous or oral cocktail of "probe drugs", depending on the route of the voriconazole dose, consisting of midazolam, ranitidine, and esomeprazole will be administered. Using the samples collected for the primary outcome, concentrations of all three probe drugs and their major metabolites will be measured and used to compute activity of the relevant drug metabolizing enzymes.

OTHER OUTCOMES:
Accuracy of computer software for Bayesian dose optimization of voriconazole in individual patients | Within 4 weeks of study completion for each subject
  Using existing voriconazole pharmacokinetic data, we have constructed a population model of the drug's behavior in children and adults. We are testing the use of this model in study subjects to compare the doses predicted by the software to achieve actual, measured voriconazole concentrations obtained for routine clinical care after the study PK visit, with the real doses that were administered and resulted in those measured voriconazole concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Neely, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Hope WW, Vanguilder M, Donnelly JP, Blijlevens NM, Bruggemann RJ, Jelliffe RW, Neely MN. Software for dosage individualization of voriconazole for immunocompromised patients. Antimicrob Agents Chemother. 2013 Apr;57(4):1888-94. doi: 10.1128/AAC.02025-12. Epub 2013 Feb 4. PMID 23380734
- [Background] Neely M, Rushing T, Kovacs A, Jelliffe R, Hoffman J. Voriconazole pharmacokinetics and pharmacodynamics in children. Clin Infect Dis. 2010 Jan 1;50(1):27-36. doi: 10.1086/648679. PMID 19951112
- [Derived] Neely M, Margol A, Fu X, van Guilder M, Bayard D, Schumitzky A, Orbach R, Liu S, Louie S, Hope W. Achieving target voriconazole concentrations more accurately in children and adolescents. Antimicrob Agents Chemother. 2015;59(6):3090-7. doi: 10.1128/AAC.00032-15. Epub 2015 Mar 16. PMID 25779580